CLINICAL TRIAL: NCT02068963
Title: Collection of Plasma and Serum Samples From Individuals Initiating Therapy With Sofosbuvir for Chronic Hepatitis C Virus Infection for the Clinical Evaluation of the Aptima HCV Quant Dx Assay
Brief Title: Collection of Plasma and Serum Samples From Individuals Initiating Sofosbuvir for Chronic Hepatitis C for Testing
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P10433-HCVQPS-01
Record Dates: First submitted 2014-02-14; First posted 2014-02-21 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Population

SUMMARY:
This non-interventional clinical study will be conducted to prospectively collect serial plasma and serum samples from treatment naïve subjects with chronic HCV infection who are initiating sofosbuvir-based therapy. These samples will be used to estimate clinical utility endpoints for the Aptima HCV Quant Dx assay which is used an aid in the management of HCV-infected patients undergoing HCV antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* The subject is chronically infected with HCV genotypes 1, 2, 3, 4, 5, and/or 6 as documented in the subject's medical records and is naïve to HCV treatment (treatment naïve).
* Chronic HCV (with or without HIV [human immunodeficiency virus] co-infection) will be documented with historical record of:
* A positive HCV RNA test result (result generated at least 6 months before the baseline visit)
* A HCV genotype test result (result generated at least 6 months before the baseline visit)
* A liver biopsy report demonstrating chronic HCV

  ---The subject is initiating antiviral therapy with a sofosbuvir regimen as indicated below:
* Sofosbuvir plus peginterferon and ribavirin for 12 weeks (peginterferon eligible genotype 1, 4, 5, or 6)
* Sofosbuvir plus ribavirin for 12 weeks (genotype 2)
* Sofosbuvir plus ribavirin for 24 weeks (peginterferon ineligible or unwilling genotype 1 or genotype 3)
* The subject is at least 18 years of age at the time of enrollment
* Adequate medical records are available for collection of protocol-defined demographics, baseline patient characteristics, medical history, virology and specific laboratory results, and other information to verify enrollment criteria
* The subject and/or legally authorized representative is willing and able to provide consent prior to providing a specimen(s)

Exclusion Criteria:

* Subjects with history or evidence of decompensated liver disease
* Subjects with severe renal impairment or end stage renal disease
* Subjects who are not naïve to HCV therapy with prior exposure to an approved or experimental HCV antiviral therapy
* Subject has characteristics that are contraindicated in the FDA approved label for sofosbuvir (eg, subjects with contraindications applicable to peginterferon and/or ribavirin, pregnant woman or men whose female partners are pregnant; Sovaldi Package Insert 2013)
* Subject is receiving treatment pre- or post-transplant
* Subject is unsuitable for study participation based on the Investigator's decision (eg, unlikely to comply with study visit schedule, significant medical complication)
* Participating in another investigational study that the Investigator believes might interfere with the subject's participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment naïve men and women ≥18 years of age with chronic HCV infection initiating sofosbuvir-based treatment will be enrolled from medical facilities that may include private and academic family practice, infectious disease, hepatology, gastroenterology, and medical group clinics.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sustained viral response based on lower limit of quantitation | 12 weeks post therapy
  Sustained viral response (SVR) is defined as viral load level being below the investigational assay's lower limit of quantitation.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kuslich, Study Director — Hologic, Inc.
Locations (34):
- United States (33):
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Franco Felizarta, MD, Bakersfield, California
  - Inland Empire Liver Foundation, Rialto, California
  - Kaiser Permanente, San Francisco, California
  - Empire Clinical Research, Upland, California
  - Island View Gastroenterology, Ventura, California
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Schiff Center for Liver Disease, Miami, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Indianapolis Gastroenterology Research Facility, Indianapolis, Indiana
  - Investigative Clinical Research, Annapolis, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Kansas City Gastroenterology, Kansas City, Missouri
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Charleston GI Specialists, Charleston, South Carolina
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Austin Center for Clinical Research, Austin, Texas
  - Cure C Consortium, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Infectious Diseases Associates of Central Virginia, Lynchburg, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - University of Washington, Seattle, Washington
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico